CLINICAL TRIAL: NCT00520533
Title: A Pilot Study of the Safety, Efficacy, and Effects on Functional Imaging of the Combination of cG250 and Sunitinib in Patients With Advanced Renal Cell Carcinoma
Brief Title: Study of Safety and Functional Imaging of cG250 and Sunitinib in Patients With Advanced Renal Cell Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed prematurely due to toxicity
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Pfizer (Industry); Heidelberg Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2007-004
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Renal Cell Carcinoma (RCC)
Keywords: Clinical trials; cG250 mAb; monoclonal antibody (mAb) G250; sunitinib; angiogenesis inhibitors; Positron-Emission Tomography; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Carcinoma, Renal Cell; Mycobacterium Infections, Nontuberculous | interventions — G250 monoclonal antibody; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- On Study (Experimental): Treatment (cycle 1):
  * cG250 10mg/m² IV weekly x 5 doses (1st & 5th doses trace-labelled with 124I)
  * Sunitinib 50 mg/day orally x 4 weeks commencing day 8
  * Followed by two-week break
  Treatment (cycle 2 - investigator discretion):
  * cG250 10mg/m² IV weekly x4 doses
  * Sunitinib 50 mg/day orally x 4 weeks (commencing concurrently)
  * Followed by two-week break
  Interventions: Biological: Chimeric monoclonal antibody cG250; Drug: Sunitinib malate

INTERVENTIONS:
Biological: Chimeric monoclonal antibody cG250 — First Cycle: cG250 10 mg/m² intravenous infusion, weekly for five weeks, followed by a two-week break. 1st & 5th dose will be trace-labeled with a radioactive substance detectable on a PET scanner (124I-cG250).
  Second cycle (investigator discretion): cG250 10 mg/m² intravenous infusion, weekly for four weeks followed by a two-week break. No 124I-cG250 will be used in the 2nd cycle.
  Up to 2 cycles available.
Drug: Sunitinib malate — First Cycle: Sunitinib 50 mg orally daily for 4 weeks (starts 8th day of 1st treatment cycle), followed by a two-week period off sunitinib.
  Second cycle (investigator discretion): Sunitinib 50 mg orally daily for 4 weeks (starts on 1st day of 2nd treatment cycle), followed by a two-week period off sunitinib.
  Up to 2 cycles available on-study.
  Other Names: Sutent

SUMMARY:
This clinical trial explores the safety, efficacy, and effects on functional imaging of cG250 monoclonal antibody (mAb) administered intravenously weekly in combination with daily oral sunitinib, in patients with advanced renal cell carcinoma.

DETAILED DESCRIPTION:
This study explores the safety, efficacy and effects on functional imaging of the combination of cG250 and sunitinib in patients with advanced renal cell carcinoma (kidney cancer).

When kidney cancer has spread beyond the kidney, it is usually not possible to cure it with surgery. Other treatments such as radiotherapy or chemotherapy are also of limited value. Kidney cancers often rely on certain proteins for their growth, particularly proteins that affect the ways that blood vessels grow into the cancer. Ingrowth of blood vessels supplies cancer cells with oxygen and nutrition; without the blood vessels, cancer deposits can not grow in size. When growth of the blood vessels is blocked, established cancers may stop growing or may shrink. This has been shown to work for some drugs that target this process in kidney cancers. One of these drugs is called sunitinib.

A protein, called G250, is also thought to be important in helping kidney cancers to grow. G250 is found on the cell surface of many kidney cancers. One possible method of interfering with the function of G250 is to target G250 with an antibody known as cG250. Clinical trials with cG250 have shown it to be safe, to home in on kidney cancer cells, and to persist in the blood and the cancer tissue for a long period of time.

The main purpose of this study is to explore whether the combination of sunitinib and cG250 is safe in patients with advanced kidney cancer. The study will also assess whether this combination is able to cause kidney cancer to shrink; will determine where cG250 travels within the body, whether the immune system reacts to the cG250 and whether sunitinib affects that; and whether the combination affects how kidney cancers grow or how blood flows within the tumour.

Eligible patients will receive cG250 10 mg/m² by weekly intravenous infusion for five weeks, followed by a two-week break (one cycle). The first and fifth dose will be trace-labeled with a radioactive substance (124I-cG250) detectable by a special scan called a Positron Emission Tomography (PET scan) to allow studies of the distribution of cG250. Sunitinib 50 mg by daily oral dose will also be given for 4 weeks (commencing on day 8 of the first treatment cycle), followed by a two-week break. Up to two cycles of treatment will be given. If a second cycle is given, cG250 will be given as four weekly doses and daily sunitinib will start on the same day. No 124I-cG250 will be administered after the first treatment cycle.

The extent of the kidney cancer will be assessed by Computed tomography (CT) at baseline and at the end of each treatment cycle. Safety assessments (physical examination, blood tests, gated cardiac blood pool scan, ECG-heart trace) will be performed at the beginning of each treatment cycle, repeated throughout the cycle and end of study. A number of blood tests and PET scans will be done in the first cycle to show how and in what amounts the 124I-cG250 distributes in the body. Other PET scans (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose {[18]F-FDG}) and 15O-water {[15]O-H2O}) will be performed to allow assessment of tumour growth and blood flow. Blood tests will also show whether the immune system recognises the infused cG250 by making an antibody against it.

A total of 14 patients were expected to be recruited; 8 were consented and 6 received study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or unresectable Renal Cell Cancer (with clear cell component).
* Measurable disease by RECIST on CT with at least one measurable lesion 2 cm or greater in diameter, which is deemed to be assessable by PET imaging.
* At least 4 weeks after chemotherapy, radiotherapy or immunotherapy (6 weeks for nitrosourea drugs).
* Expected survival at least 3 months.
* Karnofsky performance status (KPS) of 70% or greater.
* Age 18 years or older.
* Vital laboratory parameters within normal, or protocol specified ranges.
* Left ventricular ejection fraction greater than 55% on GCBP scan.
* Systolic blood pressure ≤150mmHg and diastolic blood pressure ≤90mmHg.
* Able to give written informed consent.

Exclusion Criteria:

* Prior exposure to cG250 monoclonal antibody (exception: no circulating human anti-chimeric antibody to cG250).
* Prior treatment with vascular endothelial growth factor (VEGF)-targeting agents (e.g. bevacizumab) or multi-kinase inhibitors (e.g. sorafenib) not including sunitinib. (Patients currently receiving sunitinib may be eligible if tolerating a stable dose of sunitinib on a four week on / two week off regimen, with toxicity due to sunitinib ≤ CTCAE grade 2; and for whom the investigator deems it clinically reasonable to withhold sunitinib for at least four weeks prior to commencement of study treatment.)
* Active central nervous system (CNS) metastases (exception: CNS metastases adequately treated (surgery or radiotherapy) with no progression for at least three months).
* Known HIV positivity.
* Clinically significant heart disease.
* History of hypertension requiring hospitalisation.
* Other serious illnesses, eg, serious infections requiring antibiotics, bleeding disorders.
* Major surgery or radiation therapy within 4 weeks prior to, or planned within 6 weeks of starting the study treatment. (Prior palliative radiotherapy to metastatic lesion(s) permitted, provided at least one measurable lesion was not irradiated or has progressed following radiotherapy.)
* Severe haemorrhage within 4 weeks prior to starting the study treatment.
* Any of the following within the 12 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Pre-existing thyroid abnormality with unstable thyroid function despite medication.
* Ongoing moderate to severe cardiac dysrhythmias, any severity of atrial fibrillation, or prolongation of the corrected QT interval (QTc) to greater than 450 millisecond for males or 470 millisecond for females.
* Participation in a clinical trial involving another investigational agent within 4 weeks.
* Pregnancy or breastfeeding.
* Women of childbearing potential not using a medically acceptable means of contraception.
* Psychiatric or addictive disorders that may compromise the ability to give informed consent.
* Not available for follow-up assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Ian D Davis, FRACP, FAChPM, MBBS, PhD, Principal Investigator — Ludwig Institute for Cancer Research
Locations (1):
- Austin Health (Ludwig Institute Oncology Unit), Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young H, Baum R, Cremerius U, Herholz K, Hoekstra O, Lammertsma AA, Pruim J, Price P. Measurement of clinical and subclinical tumour response using [18F]-fluorodeoxyglucose and positron emission tomography: review and 1999 EORTC recommendations. European Organization for Research and Treatment of Cancer (EORTC) PET Study Group. Eur J Cancer. 1999 Dec;35(13):1773-82. doi: 10.1016/s0959-8049(99)00229-4. PMID 10673991
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8 patients were recruited and signed informed consent; 2 patients were withdrawn prior to receiving study treatment. (One patient was withdrawn from the study because of requiring urgent radiotherapy and the other withdrew consent.) Six patients were enrolled and received study treatment.
  The study was terminated for safety reasons.
Groups:
- cG250 + Sunitinib: Treatment (cycle 1):
  * cG250 10mg/m² IV weekly x 5 doses (1st & 5th doses trace-labelled with 124I)
  * Sunitinib 50 mg/day orally x 4 weeks commencing day 8
  * Followed by two-week break
  Treatment (cycle 2 - investigator discretion):
  * cG250 10mg/m² IV weekly x4 doses
  * Sunitinib 50 mg/day orally x 4 weeks (commencing concurrently)
  * Followed by two-week break
  Up to 2 cycles available on-study.
Period: Overall Study
Arm/Group | cG250 + Sunitinib
Started | 8
Completed | 4
Not Completed | 4
Not completed — Death | 1
Not completed — Suspension of the study for safety reasons | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of cG250.
Arm/Group | cG250 + Sunitinib
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.913)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Australia | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs), Serious Adverse Events (SAEs), Dose Limiting Toxicities (DLTs) or Adverse Events Leading to Discontinuation.
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0. Adverse events (AEs) were reported based on clinical laboratory tests, vital sign, weight measurements, physical examinations, and performance status evaluations. Pre-existing symptoms were collected from the signing of informed consent until the first dose of study drug. Adverse events were collected from the first dose of study drug through the end of study assessment.
  Dose Limiting Toxicity (DLT): any of the following events occurring within 30 days of study drug administration related to cG250 or sunitinib.
  Grade 2 or greater allergic reaction. Grade 3 toxicity. Exceptions are: fever; asymptomatic hyperglycemia; hypophosphatemia; nausea, vomiting, or diarrhoea that resolve with medical therapy; leukopenia or thrombocytopenia that revert to baseline within three weeks of occurrence, or lymphopenia only.
  Any Grade 4 toxicity.
Time Frame: up to 14 weeks
Population: All patients who received at least one dose of cG250.
Measure: Count of Participants; unit: Participants
Groups:
- cG250 and Sunitinib: Treatment (cycle 1):
  * cG250 10mg/m² IV weekly x 5 doses (1st & 5th doses trace-labelled with 124I)
  * Sunitinib 50 mg/day orally x 4 weeks commencing day 8
  * Followed by two-week break
  Treatment (cycle 2 - investigator discretion):
  * cG250 10mg/m² IV weekly x4 doses
  * Sunitinib 50 mg/day orally x 4 weeks (commencing concurrently)
  * Followed by two-week break
  Up to 2 cycles available on-study.
Arm/Group | cG250 and Sunitinib
Number analyzed (Participants) | 6
Participants
  Number of Patients With at least 1 AE | 6
  Number of Patients With at Least 1 Serious AE | 3
  Number of Patients With a DLT | 2
  Number of Patients with an AE leading to treatment discontinuation | 1

2. Secondary Outcome: Number of Patients With Tumour Response Assessed by Response Evaluation Criteria in Solid Tumors (RECIST).
Description: Tumor responses were evaluated using appropriate imaging and categorized according to RECIST at Screening (within 4 weeks of the first dose of study treatment), and after cycles 1 and 2 of study treatment. Per RECIST, target lesions are categorized as follows: complete response (CR): disappearance of all target lesions; partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; progressive disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria (Therasse et al 2000).
Time Frame: up to 14 weeks
Population: All patients who received at least one dose of cG250.and were evaluable for tumour response.
Measure: Count of Participants; unit: Participants
Arm/Group | cG250 + Sunitinib
Number analyzed (Participants) | 4
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 1
  Stable Disease (SD) | 3
  Progressive Disease (PD) | 0

3. Secondary Outcome: Number of Patients With Tumor Metabolic Response as Assessed by Serial 18F-FDG-PET Scans.
Description: 18F-FDG-PET was performed at pre-study, between days 15-22 and at the end of cycle 1. At baseline, visual grading of the intensity of FDG uptake was scored. On follow-up PET scans, the greatest baseline maximum standard uptake value (SUVmax) of the reference lesion with the greatest baseline value and presence/absence of new sites of disease were recorded.
  Tumour metabolic response was calculated using the SUVmax and was categorized according to the EORTC guidelines (Young et al 1999).
  Complete metabolic remission (CMR) is the disappearance of tracer uptake in the target lesion and no new lesions; Partial metabolic remission (PMR) is a 20% or more decrease in the tracer uptake in the target lesion and no new lesions; Tumor progression was defined as a greater than 20% increase in FDG uptake or the appearance of new tumour lesions. Stable metabolic disease (SMD) was classified as no significant change in uptake.
Time Frame: 7 weeks
Population: All patients who received at least one dose of cG250, completed cycle 1 and were evaluable for tumor metabolic response.
Measure: Count of Participants; unit: Participants
Arm/Group | cG250 + Sunitinib
Number analyzed (Participants) | 4
Participants
  CMR | 1
  PMR | 0
  SMD | 3

4. Secondary Outcome: Whole Body Clearance as Measured by Mean Biological Half-life (T1/2) After the First and Fifth Infusions of 124I-cG250.
Description: Biological half-life is the clearance of the 124I from the whole body. Positron emission tomography (PET) imaging was performed at 1 - 4 hours post infusion, and at two other time points over the ensuing one-week period.
  Quantitative uptakes of 124I-cG250 were assessed in one selected reference tumour lesion identified by 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (18F-FDG) PET imaging. Tumour volume of Interest (VOI) was delineated around the whole tumour mass on the consecutive transverse slices of FDG-PET/CT images at which the tumours were most clearly identified.
  Whole body clearance of 124I-cG250 was calculated from the whole body PET volumetric images, obtained at the multiple imaging time points after infusion. VOIs were delineated to encompass the whole body regions in the images, and for the whole-body VOI at each time point, the total counts per minute was normalized to the first imaging time point on Day 1.
Time Frame: 7 weeks
Population: All patients who received the first and fifth infusion of 124I-cG250. Two patients received the first infusion but not the fifth infusion and as a result were not included in the Week 5 results.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | cG250 + Sunitinib
Number analyzed (Participants) | 6
days
  Biological T1/2 Week 1 | 121.12 (20.68)
  Biological T1/2 Week 5: number analyzed (Participants) | 4
  Biological T1/2 Week 5 | 149.12 (42.52)
Statistical Analysis 1: Comparison: cG250 + Sunitinib; Comparison of Biological T1/2 at Week 1 and Week 5; Test type: Superiority; p = 0.194, t-test, 2 sided

5. Secondary Outcome: Whole Body Clearance as Measured by Mean Effective Half-life (T1/2) After the First and Fifth Infusions of 124I-cG250.
Description: Effective half-life is the time it takes the radiolabel to be reduced by 50%. This takes into account the biological elimination and the radioactive decay of the 124I.
  PET imaging studies were performed at 1 - 4 hours post infusion, and at two other time points over the ensuing one-week period.
  Quantitative uptakes of 124I-cG250 were assessed in one selected reference tumour lesion identified by 18F-FDG-PET imaging. Tumour volume of Interest (VOI) was delineated around the whole tumour mass on the consecutive transverse slices of FDG-PET/CT images at which the tumours were most clearly identified.
  Whole body clearance of 124I-cG250 was calculated from the whole body PET volumetric images, obtained at the multiple imaging time points after infusion. VOIs were delineated to encompass the whole body regions in the images, and for the whole-body VOI at each time point, the total counts per minute was normalized to the first imaging time point on Day 1.
Time Frame: 7 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | cG250 + Sunitinib
Number analyzed (Participants) | 6
hours
  Effective T1/2 Week 1 | 54.46 (5.00)
  Effective T1/2 Week 5: number analyzed (Participants) | 4
  Effective T1/2 Week 5 | 59.15 (6.40)
Statistical Analysis 1: Comparison: cG250 + Sunitinib; Comparison of Effective T1/2 at Week 1 and Week 5; Test type: Superiority; p = 0.172, t-test, 2 sided

6. Secondary Outcome: Number of Patients With 124I-cG250 Tumor Uptake After the First and Fifth Infusions of 124I-cG250.
Description: PET imaging studies were performed at 1 - 4 hours post infusion, and at two other time points over the ensuing one-week period.
  Quantitative uptakes of 124I-cG250 were assessed in one selected reference tumour lesion identified by 18F-FDG-PET imaging. Tumour volume of Interest (VOI) was delineated around the whole tumour mass on the consecutive transverse slices of FDG-PET/CT images at which the tumours were most clearly identified.
  Uptakes of 124I-cG250 were assessed in one selected reference tumour lesion identified by 18F-FDG-PET imaging.
Time Frame: 7 weeks
Population: All patients who received the first and fifth infusion of 124I-cG250. Two patients received the first infusion but not the fifth infusion and as a result were not included in the tumour uptake after the fifth infusion of 124I-cG250.
Measure: Count of Participants; unit: Participants
Arm/Group | cG250 + Sunitinib
Number analyzed (Participants) | 6
Participants
  First Infusion: Tumor uptake | 6
  First Infusion: No Tumor uptake | 0
  Fifth Infusion: number analyzed (Participants) | 4
  Fifth Infusion: Tumor uptake | 4
  Fifth Infusion: No Tumor uptake | 0

7. Secondary Outcome: Serum Pharmacokinetics as Measured by Mean Initial Half-life (T½ α) and Mean Terminal Half-life (T½ β) After the First and Fifth Infusions of 124I-cG250 as Measured by Blood 124I Radioactivity and After the First Dose as Measured by ELISA.
Description: Blood samples were taken prior to 124I-cG250 infusion and 5 minutes, 1, 2, 4 and 24 hours post 124I-cG250 infusion. The pharmacokinetics of 124I-cG250 were calculated using gamma scintillation counting and by enzyme-linked immunosorbent assay (ELISA).
Time Frame: 7 weeks
Population: All patients who received the first and fifth infusion of 124I-cG250. Two patients received the first infusion but not the fifth infusion and as a result were not included in the fifth infusion results. Two patients were not included in the T½ β ELISA analysis due to a disproportionate effect on the estimated parameter.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | cG250 + Sunitinib
Number analyzed (Participants) | 6
hours
  T½ α as measured by blood 124I radioactivity after the first infusion | 9.83 (8.63)
  T½ β as measured by blood 124I radioactivity after the first infusion | 104.1 (52.2)
  T½α as measured by ELISA after the first infusion | 27.7 (34.4)
  T½ β as measured by ELISA after the first infusion: number analyzed (Participants) | 4
  T½ β as measured by ELISA after the first infusion | 105.2 (52.2)
  T½ α as measured by blood 124I radioactivity after the fifth infusion: number analyzed (Participants) | 4
  T½ α as measured by blood 124I radioactivity after the fifth infusion | 18.54 (14.04)
  T½ β as measured by blood 124I radioactivity after the fifth infusion: number analyzed (Participants) | 4
  T½ β as measured by blood 124I radioactivity after the fifth infusion | 146.9 (69.2)

8. Secondary Outcome: Serum Pharmacokinetics as Measured by Mean Volume of Central Compartment (V1) After the First and Fifth Infusions of 124I-cG250 as Measured by Blood 124I Radioactivity and After the First Dose as Measured by ELISA.
Description: as for outcome 7
Time Frame: 7 weeks
Population: All patients who received the first and fifth infusion of 124I-cG250. Two patients received the first infusion but not the fifth infusion and as a result were not included in the fifth infusion results.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | cG250 + Sunitinib
Number analyzed (Participants) | 6
mL
  V1 as measured by blood 124I radioactivity after the first infusion | 3067 (705)
  V1 as measured by blood 124I radioactivity after the fifith infusion: number analyzed (Participants) | 4
  V1 as measured by blood 124I radioactivity after the fifith infusion | 2542 (267)
  V1 as measured by ELISA after the first infusion | 2286 (678)

9. Secondary Outcome: Serum Pharmacokinetics as Measured by Mean Area Under the Concentration Curve Extrapolated to Infinite Time (AUC) After the First and Fifth Infusions of 124I-cG250 as Measured by Blood 124I Radioactivity and After the First Dose as Measured by ELISA.
Description: as for outcome 7
Time Frame: 7 weeks
Population: All patients who received the first and fifth infusion of 124I-cG250. Two patients received the first infusion but not the fifth infusion and as a result were not included the fifth infusion results. Two patients were not included in the ELISA analysis due to a disproportionate effect on the estimated parameter.
Measure: Mean (Standard Deviation); unit: hours*mcg/mL
Arm/Group | cG250 + Sunitinib
Number analyzed (Participants) | 6
hours*mcg/mL
  AUC as measured by blood 124I radioactivity after the first infusion | 520 (153)
  AUC as measured by blood 124I radioactivity after the fifth infusion: number analyzed (Participants) | 4
  AUC as measured by blood 124I radioactivity after the fifth infusion | 682 (240)
  AUC as measured by ELISA after the first infusion: number analyzed (Participants) | 4
  AUC as measured by ELISA after the first infusion | 759 (335)

10. Secondary Outcome: Serum Pharmacokinetics as Measured by Mean Total Serum Clearance (CL) After the First and Fifth Infusions of 124I-cG250 as Measured by Blood 124I Radioactivity and After the First Dose as Measured by ELISA.
Description: as for outcome 7
Time Frame: 7 weeks
Population: All patients who received the first and fifth infusion of 124I-cG250. Two patients received the first infusion but not the fifth infusion and as a result were not included in the fifth infusion results. Two patients were not included in the ELISA analysis due to a disproportionate effect on the estimated parameter.
Measure: Mean (Standard Deviation); unit: mL/hour
Arm/Group | cG250 + Sunitinib
Number analyzed (Participants) | 6
mL/hour
  CL as measured by blood 124I radioactivity after the first infusion | 38.7 (19.7)
  CL as measured by blood 124I radioactivity after the fifth infusion: number analyzed (Participants) | 4
  CL as measured by blood 124I radioactivity after the fifth infusion | 28.7 (15.7)
  CL as measured by ELISA after the first infusion: number analyzed (Participants) | 4
  CL as measured by ELISA after the first infusion | 25.7 (17.5)

11. Secondary Outcome: Serum Pharmacokinetics as Measured by Mean Maximum Serum Concentration (Cmax) After the First and Fifth Infusions of 124I-cG250 as Measured by Blood 124I Radioactivity and After the First Dose as Measured by ELISA.
Description: as for outcome 7
Time Frame: 7 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | cG250 + Sunitinib
Number analyzed (Participants) | 6
mcg/mL
  Cmax as measured by blood 124I radioactivity after the first infusion | 5.93 (1.06)
  Cmax as measured by blood 124I radioactivity after the fifth infusion: number analyzed (Participants) | 4
  Cmax as measured by blood 124I radioactivity after the fifth infusion | 6.661 (0.678)
  Cmax as measured by ELISA after the first infusion | 7.57 (1.88)

12. Secondary Outcome: Number of Patients With Decreases in Tumour Blood Flow on Week 3 Versus Baseline.
Description: 15O-H2O PET scans were performed up to 14 days prior to treatment and between days 15-22 in the first treatment cycle only. Approximately 750 megabecquerel (MBq) of 15O-H2O were administered intravenously and data was acquired dynamically over 5-10 minutes. The PET scan field of view was of an anatomical region containing a least one reference tumour lesion. Quantitation of blood flow within tumour was performed, and expressed in mL/mg/min. Follow-up 15O-H2O PET scan quantitated blood flow within the same reference lesion(s), allowing direct comparison of any change in quantitative tumour blood flow in response to treatment to be measured.
Time Frame: 7 weeks
Population: Number of patients who received 15O-H2O PET scans at baseline and between days 15-22. One patient did not receive the 15O-H2O PET scans due to technical problems.
Measure: Count of Participants; unit: Participants
Arm/Group | cG250 + Sunitinib
Number analyzed (Participants) | 5
Participants | 5

13. Secondary Outcome: Number of Patients With Human Anti-chimeric Antibodies (HACA)
Description: Blood samples (5 mL/sample) were drawn prior to each cG250 or 124I-cG250 infusion during cycle 1 and also at the End of Study visit. If a second cycle of treatment was administered, HACA was performed at the End of Study visit.
  The immunochemical measurement of anti-cG250 antibodies in human serum was performed by an enzyme-linked immunosorbent assay (ELISA).
  Samples with values greater than the limit of quantitation (16 ng/mL) were considered HACA positive. Samples at or below that level were reported as negative.
Time Frame: 7 - 14 weeks
Population: All patients who had one cG250 pre-treatment and at least one post-treatment sample taken.
Measure: Count of Participants; unit: Participants
Arm/Group | cG250 + Sunitinib
Number analyzed (Participants) | 6
Participants
  Number of patients with positive HACA | 0
  Number of patients with negative HACA | 6

ADVERSE EVENTS:
Time Frame: up to 14 weeks
Description: Toxicity will be evaluated according to the National Cancer Institute CTCAE Scale (Version 3.0).
  All events, which occurred after signed informed consent, but before first administration of study drug, were documented on the Pre-existing Signs and Symptom page. Thereafter, they were documented on the Adverse Event page.
Arm/Group | cG250 + Sunitinib
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | cG250 + Sunitinib (N=6)
Vomiting (Gastrointestinal disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Left pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | cG250 + Sunitinib (N=6)
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Pharyngitis (Infections and infestations) | 1
Blood creatinine increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 3
Skin discoloration (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Ventricular ectopics (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hazy vision (Eye disorders) | 1
Visual disturbance (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Facial swelling (Skin and subcutaneous tissue disorders) | 1
Loose Tooth (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Tooth abscess (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Tenth rib fracture (Injury, poisoning and procedural complications) | 1
GFR decreased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Leg pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Dysphasia (Nervous system disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Insomnia (Psychiatric disorders) | 2
Balanitis (Reproductive system and breast disorders) | 1
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Lightheadedness (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Tremor of hands (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No